CLINICAL TRIAL: NCT00828737
Title: Prospective Non-randomized (Pharmacoepidemiologic) Cohort Study (Open-label, Multicenter) to Assess the Magnitude of Potential Risk With the Administration of Gadovist in Patients With Moderate to Severe Renal Impairment for the Development of Nephrogenic Systemic Fibrosis (NSF) Based on Diagnostically Specific Clinical and Histopathologic Information
Brief Title: Safety of Gadovist in Renally Impaired Patients
Acronym: GRIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13273; 2008-004496-22 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2009-01-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Fibrosis; Renal Impairment
MeSH Terms: conditions — Fibrosis; Renal Insufficiency | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — Gadovist in approved indications at approved dosages

SUMMARY:
Patients with moderate to severe renal impairment scheduled for a magnetic resonance imaging (MRI) scan and injection with a contrast agent, Gadovist, will be asked to participate.

The administration of contrast agents that contain gadolinium such as Gadovist might increase a potential risk to develop a rare condition called nephrogenic systemic fibrosis (NSF) in patients with renal impairment. This study is to assess the potential risk to develop NSF in patients with renal impairment after the administration of Gadovist. Patients who are enrolled in this study will receive a Gadovist enhanced MRI scan which was prescribed by the referring doctor. After the MRI scan the patient will be included in a two year follow-up period to assess if signs or symptoms suggestive of NSF have appeared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate (eGFR 30 - 59 ml/min/173m2) or severe (eGFR < 30 ml/min/1.73m2) renal impairment, scheduled to undergo Gadovist-enhanced MRI

Exclusion Criteria:

* GBCA-enhanced MRI (or administration of a GBCA for any other CE imaging procedure) other than Gadovist within 12 months prior to administration of Gadovist
* History of NSF (Nephrogenic Fibrosing Dermopathy)
* Age outside the indicated age range mentioned in national labelling.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2008-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with moderate to severe renal impairment, who develop Nephrogenic Systemic Fibrosis (NSF), based on diagnostically specific clinical and histopathological information | From the time of MRI until the end of follow-up period (24 months)

SECONDARY OUTCOMES:
Number of Participants With Moderate to Severe Renal Impairment in Whom no Biopsy was Obtained who Develop Nephrogenic Systemic Fibrosis (NSF) Based on Diagnostically Specific Clinical Information | From the time of MRI until the end of follow-up period (24 months)
Number of Participants With Different Criteria of Diagnostic Confidence of the Investigator Based on | Immediately after Gadovist-enhanced MRI
Number of Participants With Image Quality Sufficient for Diagnosis | Immediately after Gadovist-enhanced MRI
Evaluation of Creactive Protein (CRP) in Participants With Moderate and Severe Renal Impairment | Within 48 hours prior to the Gadovist administration
Evaluation of Macrophage Inflammatory Proteins (MIP) and Monocyte Chemotactic Proteins (MCP) in Participants With Moderate and Severe Renal Impairment | Within 48 hours prior to the Gadovist administration
Evaluation of Osteopontin and Tissue Inhibitor of Metallo Proteinase 1 (TIMP1) in Participants With Moderate and Severe Renal Impairment | Within 48 hours prior to the Gadovist administration
Number of Participants With Treatmentemergent Adverse Events (TEAEs), Treatmentemergent Serious Adverse Event (TESAE), Drugrelated Treatmentemergent Adverse Events (TEAEs) and Drugrelated Treatmentemergent Serious Adverse Events (TESAEs) | From the time of MRI until the end of follow-up period (24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (61):
- Australia (4):
  - Adelaide, South Australia
  - Clayton, Victoria
  - Geelong, Victoria
  - Westmead NSW
- Austria (5):
  - Innsbruck, Tyrol
  - Ehenbichl
  - Graz
  - Leoben
  - Vienna
- Canada (4):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Toronto, Ontario
  - Fleurimont, Quebec
- France (5):
  - Le Kremlin-Bicêtre
  - Lille
  - Marseille
  - Paris
  - Reims
- Germany (19):
  - Mannheim, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Coburg, Bavaria
  - Erlangen, Bavaria
  - München, Bavaria
  - Regensburg, Bavaria
  - Neuruppin, Brandenburg
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Hannoversch Münden, Lower Saxony
  - Osnabrück, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Lüdenscheid, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia
- Italy (12):
  - Rozzano, Milano
  - Ancona
  - Brescia
  - Florence
  - Genova
  - Milan
  - Napoli
  - Pisa
  - Roma
  - Torino
  - Treviso
  - Verona
- South Korea (5):
  - Seongnam-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Jeonju-Si, Jeonrabuk-Do
  - Seoul
- Spain (3):
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Granada, Granada
- Switzerland (2):
  - Basel, Canton of Basel-City
  - Lugano, Canton Ticino
- Thailand (2):
  - Bangkok
  - Songkhla

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/